CLINICAL TRIAL: NCT00100932
Title: Phase II Study of E7389, a Halichondrin B Analog, in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC), Who Progressed During or After Platinum-Based Doublet Chemotherapy Stratified for Prior Taxane Therapy
Brief Title: Phase II Study Of E7389, Halichondrin B Analogue, In Patients With Advanced Non-Small Cell Lung Cancer, NSCLC, Who Progressed During Or After Platinum-Based Doublet Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7389-A001-202
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Results first posted 2012-01-31 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Non-Small-Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — eribulin

ARMS (2):
- 1 (Experimental): E7389 28 day cycle
  Interventions: Drug: E7389 28 Day Cycle
- 2 (Experimental): E7389 21 day cycle
  Interventions: Drug: E7389 21 Day Cycle

INTERVENTIONS:
Drug: E7389 28 Day Cycle — E7389 1.4 mg/m^2 IV bolus on Days 1, 8, and 15 of a 28 day cycle.
  Arms: 1
Drug: E7389 21 Day Cycle — E7389 1.4 mg/m^2 IV bolus on Days 1 and 8 of a 21 day cycle.
  Arms: 2

SUMMARY:
This is a study of E7389 in patients with recurrent and/or metastatic Non-Small-Cell Lung Cancer (NSCLC) who progressed during or after treatment with a platinum agent and another chemotherapy.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients must have a histologically or cytologically confirmed diagnosis of non-small cell lung cancer with at least one site of measurable disease by the RECIST criteria.
* Patients must have failed prior platinum-containing doublet chemotherapy. Patients who have received single agent chemotherapy with or without a subsequent taxane containing regimen may be enrolled after discussion with Sponsor.
* Patients must be ≥ 18 years of age.
* Patients must have a performance score of 0 or 1 using the ECOG performance scale.
* Patients must have a life expectancy of ≥ 3 months.
* Patients must have adequate renal function as evidenced by a serum creatinine ≤ 2.0 mg/dL or a calculated creatinine clearance ≥ 40 mL/min per the Cockcroft and Gault formula.
* Patients must have adequate hepatic function as evidenced by bilirubin ≤1.5 mg/dL and alkaline phosphatase, AST and ALT ≤ 3 times upper limit of normal, unless there is evidence of liver metastases, in which case the alkaline phosphatase, AST and ALT must be ≤ 5 times upper limit of normal.
* Patients must have adequate bone marrow function as evidenced by absolute neutrophil counts (ANC) ≥ 1.5 X 10^9/L, hemoglobin ≥ 10.0 g/dL (a hemoglobin < 10.0 g/dL would be acceptable if it can be corrected by growth factor or transfusion), and platelet count ≥ 100 X 10^9/L.
* Patients must be willing and able to comply with the protocol guidelines for the duration of the study.
* Patients must be willing and able to complete the Lung Cancer Symptom Scale (LCSS) instrument.
* The biopsy specimen (paraffin block or at least 10 unstained slides) must be available from either the initial diagnosis or any subsequent diagnostic or surgical procedure of patients participating in the pharmacogenomics sub-study only. However, no additional biopsies are obligatory for participation in this study except those required for confirmation of the diagnosis.
* Patients must give written informed consent prior to any study-specific screening procedures with the understanding that the patient may withdraw consent at any time without prejudice.

EXCLUSION CRITERIA:

* Patients with pre-existing peripheral neuropathy > Grade 2
* Patients who require therapeutic doses of warfarin
* Patients who have not recovered from any chemotherapy, radiation or other therapy related toxicity deemed to be clinically significant at study entry
* Patients with active symptomatic brain metastases. Patients with central nervous system (CNS) metastases are considered eligible if they have had adequately treated brain metastases, i.e. have completed treatment (tapered off steroids) at least four weeks before starting treatment with E7389. Patients who have no evidence that the metastases are symptomatic or actively growing (no evidence of midline shift on CT scan or MRI) may be enrolled without initiation of local therapy for the CNS metastases. In this case, a repeat scan must be performed within four weeks of the original scan to ensure that disease progression is not occurring. It is not the intention of this study to treat patients with active brain metastases.
* Patients who have a positive history for HIV, active hepatitis B or active hepatitis C.
* Patients with other significant medical, or psychiatric disorders that, in the opinion of the investigator, will exclude the patient from the study for compliance or safety reasons
* Patients who have received investigational drugs, including immunotherapy, gene therapy, hormone therapy (except megestrol acetate for appetite stimulation), or other biological therapy; conventional chemotherapy or radiation therapy (except for palliation, defined as less than 10% of the bone marrow reserve and less than 20 Gy), within three weeks of E7839 enrollment
* Patients who have received non-cytotoxics (eg, gefitinib, erlotinib) within one week of E7389 enrollment
* Patients who have not recovered from major surgery within three weeks of E7389 enrollment
* Patients with severe/uncontrolled intercurrent illness/infection
* Patients with significant cardiovascular impairment (history of congestive heart failure>NYHA grade II, unstable angina or myocardial infarction within the past six months, or serious cardiac arrhythmia)
* Patients with organ allografts
* Patients with hypersensitivity to halichondrin B and/or halichondrin B-related compounds
* Patients who participated in a prior E7389 clinical trial
* Patients with second malignancy within the past 5 years, except for carcinoma in situ of the cervix or basal cell carcinoma of the skin
* Women who are pregnant or breast-feeding; woman of childbearing potential with a positive pregnancy test at screening or no pregnancy test. Women of childbearing potential unless (1) surgically sterile or (2) using adequate measures of contraception in the opinion of the Investigator. Perimenopausal women must be amenorrheic for at least 12 months or using adequate contraception to be considered of non-childbearing potential.
* Fertile men who are not willing to use contraception or fertile men with a female partner who is not willing to use contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2004-12; Primary Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dale Shuster, Ph.D., Study Director — Eisai Inc.
Locations (13):
- United States (13):
  - Gilroy, California
  - Ocala, Florida
  - Baltimore, Maryland
  - Columbia, Missouri
  - Saint Joseph, Missouri
  - St Louis, Missouri
  - McCook, Nebraska
  - Canton, Ohio
  - Dallas, Texas
  - Fort Worth, Texas
  - Fairfax, Virginia
  - Norfolk, Virginia
  - Vancouver, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 29 centers in the US during the period of Dec 2004 to Apr 2006.
Groups:
- E7389 28 Day Cycle: E7389 1.4 mg/m^2 intravenous bolus on Days 1, 8 and 15 of a 28 day cycle.
- E7389 21 Day Cycle: E7389 1.4 mg/m^2 intravenous bolus on Days 1 and 8 of a 21 day cycle.
Period: Overall Study
Arm/Group | E7389 28 Day Cycle | E7389 21 Day Cycle
Started | 78 (Represents all enrolled pts; counts in demographic section represents ITT/Safety Population.) | 28 (Represents all enrolled pts; counts in demographic section represents ITT/Safety Population.)
Completed | 5 | 1
Not Completed | 73 | 27
Not completed — Adverse Event | 11 | 2
Not completed — Withdrawal by Subject | 6 | 0
Not completed — Progressive Disease | 44 | 18
Not completed — Physician Decision | 7 | 5
Not completed — Other | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E7389 28 Day Cycle | E7389 21 Day Cycle | Total
Number analyzed (Participants) | 77 | 26 | 103
Age Continuous [Mean (Standard Deviation); unit: years] | 62.0 (10.59) | 65.5 (8.97) | 62.9 (10.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 14 | 52
  Male | 39 | 12 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 75 | 26 | 101
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 1 | 8
  White | 65 | 24 | 89
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 77 | 26 | 103

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response Rate (ORR)
Description: Based on Response Evaluation Criteria in Solid Tumors (RECIST), consisting of complete response (CR) plus partial response (PR). Defined as the best response from the start of treatment until disease progression or recurrence. Lesions measured by computed tomography (CT) scan and magnetic resonance imaging (MRI). Objective response rate: complete response (CR-disappearance of all lesions)+ partial response (PR-30% decrease in lesion diameter), Progressive Disease (PD-20% increase in lesion diameter), stable disease (SD-neither shrinkage nor increase of lesions).
Time Frame: From start of treatment until disease progression or recurrence
Population: Intent to Treat/Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | E7389 28 Day Cycle | E7389 21 Day Cycle
Number analyzed (Participants) | 77 | 26
percentage of participants | 11.7 | 3.8

2. Secondary Outcome: Duration of Response
Description: Measured from the time that measurement criteria were met for complete response (CR) and partial response (PR) until the first date that recurrence or progressive disease was objectively documented.
Time Frame: From time of CR or PR until recurrence or progressive disease
Population: Intent to Treat/Safety Population
Measure: Median (Full Range); unit: Days
Arm/Group | E7389 28 Day Cycle | E7389 21 Day Cycle
Number analyzed (Participants) | 77 | 26
Days | 171 [50 to 291] | 176 [176 to 176]

3. Secondary Outcome: Progression Free Survival
Description: Defined as the time from the start of study medication until progressive disease or death from any cause during the study period.
Time Frame: From start of study medication until progressive disease or death
Population: Intent to Treat/Safety Population
Measure: Median (Full Range); unit: Days
Arm/Group | E7389 28 Day Cycle | E7389 21 Day Cycle
Number analyzed (Participants) | 77 | 26
Days | 106 [1 to 408] | 78 [1 to 218]

4. Secondary Outcome: Overall Survival
Description: Defined as the time from the start of study medication until death from any cause.
Time Frame: From time of start of study medication until death
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | E7389 28 Day Cycle | E7389 21 Day Cycle
Serious Adverse Events (participants affected / at risk) | 33/77 | 11/26
Other Adverse Events (participants affected / at risk) | 77/77 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E7389 28 Day Cycle (N=77) | E7389 21 Day Cycle (N=26)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac Tamponade (Cardiac disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
Diverticular Perforation (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Disease Progression (General disorders) | 5 | 0
Pain (General disorders) | 2 | 1
Pyrexia (General disorders) | 3 | 0
Cellulitis (Infections and infestations) | 0 | 1
Neutropenic Sepsis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 1
Pyrothorax (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Blood Pressure Systolic Inspiratory Decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Coordination Abnormal (Nervous system disorders) | 1 | 1
Dysarthria (Nervous system disorders) | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 1 | 0
Status Epilepticus (Nervous system disorders) | 1 | 0
Hallucinations, Visual (Psychiatric disorders) | 1 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Deep Vein Thrombosis (Vascular disorders) | 0 | 3
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E7389 28 Day Cycle (N=77) | E7389 21 Day Cycle (N=26)
Leukopenia (Blood and lymphatic system disorders) | 5 | 3
Neutropenia (Blood and lymphatic system disorders) | 44 | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2
Atrial Fibrillation (Cardiac disorders) | 1 | 2
Tachycardia (Cardiac disorders) | 5 | 0
Abdominal Pain (Gastrointestinal disorders) | 10 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 30 | 15
Diarrhea (Gastrointestinal disorders) | 19 | 9
Dry Mouth (Gastrointestinal disorders) | 5 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 6 | 0
Nausea (Gastrointestinal disorders) | 38 | 13
Stomatitis (Gastrointestinal disorders) | 14 | 1
Vomiting (Gastrointestinal disorders) | 24 | 6
Asthenia (General disorders) | 13 | 4
Chest Pain (General disorders) | 8 | 4
Chills (General disorders) | 7 | 14
Fatigue (General disorders) | 50 | 15
Gait Disturbance (General disorders) | 4 | 0
Mucosal Inflammation (General disorders) | 11 | 2
Edema (General disorders) | 7 | 2
Edema Peripheral (General disorders) | 15 | 7
Pain (General disorders) | 5 | 3
Pyrexia (General disorders) | 24 | 6
Bronchitis (Infections and infestations) | 1 | 2
Candidiasis (Infections and infestations) | 5 | 1
Herpes Zoster (Infections and infestations) | 1 | 3
Oral Candidiasis (Infections and infestations) | 5 | 0
Pneumonia (Infections and infestations) | 7 | 2
Sinusitis (Infections and infestations) | 8 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 10 | 5
Urinary Tract Infection (Infections and infestations) | 12 | 3
Excoriation (Injury, poisoning and procedural complications) | 4 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 2
Breath Sounds Abnormal (Investigations) | 10 | 2
Weight Decreased (Investigations) | 12 | 2
Anorexia (Metabolism and nutrition disorders) | 30 | 11
Decreased Appetite (Gastrointestinal disorders) | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 10 | 2
Hyperglycemia (Gastrointestinal disorders) | 8 | 1
Hypokalemia (Metabolism and nutrition disorders) | 5 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 6 | 2
Hyponatremia (Metabolism and nutrition disorders) | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 5
Bone Pain (Musculoskeletal and connective tissue disorders) | 11 | 4
Flank Pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 7 | 2
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 4 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 6 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 7 | 3
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Dizziness (Nervous system disorders) | 11 | 7
Dysgeusia (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 7 | 2
Hypoaesthesia (Nervous system disorders) | 5 | 2
Neuropathy (Nervous system disorders) | 11 | 4
Neuropathy Peripheral (Nervous system disorders) | 12 | 4
Paraesthesia (Nervous system disorders) | 4 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 7 | 4
Somnolence (Nervous system disorders) | 5 | 1
Anxiety (Psychiatric disorders) | 15 | 5
Confusional State (Psychiatric disorders) | 6 | 0
Depression (Psychiatric disorders) | 18 | 3
Insomnia (Psychiatric disorders) | 16 | 4
Pollakiuria (Renal and urinary disorders) | 6 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 37 | 12
Dyspnea Exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 10 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 34 | 4
Night Sweats (Skin and subcutaneous tissue disorders) | 5 | 1
Rash (Skin and subcutaneous tissue disorders) | 11 | 3
Deep Vein Thrombosis (Vascular disorders) | 1 | 3
Hypotension (Vascular disorders) | 7 | 1
Phlebitis (Vascular disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No